CLINICAL TRIAL: NCT06895590
Title: The HIgh-fidelity Hydraulic couPling Upper-arm Cuff Assessment of Limits, Safety, and Effectiveness (HIPULSE) Trial
Acronym: HIPULSE
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: BP FR_ AMC vs A-line and NIBP
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery, Non-Cardiac ICU
Keywords: BP, FR, DBP, MAP, SBP, A-line

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Philips AMC Cuff: This is a non-randomized, single arm, self-controlled observational study. The Philips AMC cuff will be tested on all enrolled participants.
  Interventions: Device: Philips Advanced Monitoring Cuff (i.e. AMC)

INTERVENTIONS:
Device: Philips Advanced Monitoring Cuff (i.e. AMC) — Investigational, non-invasive upper arm cuff

SUMMARY:
The purpose of this study is to compare measurements of blood pressure (BP) and fluid responsiveness between the Philips AMC and invasive radial arterial line in surgical patients.

DETAILED DESCRIPTION:
Primary Objective:

• To evaluate equivalence of BP measurements (Systolic Blood Pressure [SBP], Diastolic Blood Pressure [DBP], and Mean Arterial Pressure [MAP]) derived from the Philips AMC to the radial arterial line as ground truth.

Secondary Objectives:

* To evaluate equivalence of Pulse Rate (PR) obtained by the Philips AMC to the radial arterial line as the ground truth.
* To evaluate equivalence of Pulse Pressure Variation (PPV) obtained by the Philips AMC to calculated PPV obtained using the radial arterial line waveform pulse pressures as the ground truth.
* To evaluate equivalence of Stroke Volume Variation (SVV) obtained by the Philips AMC to calculated SVV (e.g. from a predicate device that uses the radial arterial line waveform) as the ground truth.
* To evaluate superiority of blood pressure measurements obtained by the Philips AMC to the oscillometric non-invasive blood pressure (NIBP) cuff, with the radial arterial line as the reference.
* To evaluate trending agreement of BP and fluid responsiveness measurements.
* To assess time to apply the Philips AMC relative to the radial arterial line.
* To assess time from set-up start to first measurement completion between the Philips AMC and radial arterial line.
* To collect and report safety data from the Philips AMC.
* To collect and report system user experience and satisfaction scores from Philips AMC users.
* To create a research dataset with the collected data to use for future hemodynamic algorithm development and validation.

Hypothesis: Blood pressure measurements derived from the Philips AMC are equivalent to the radial arterial line and superior to the oscillometric non-invasive blood pressure (NIBP) cuff.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Indication for NIBP cuff
* Indication for a radial arterial line
* Subject or legal authorized representative is able to understand and speak the local language (also Spanish for US sites) to provide voluntary written informed consent prior to study procedures

The following stratification criteria must be met across the study sites and hence targeted enrollment may be required:

* Age of every patient 18+; at least 30% > 65 years, 30% ≤ 65 years
* At least 30% male, 30% female
* Minimum number of subjects needed to test each size cuff (per ISO81060-2:2018/AMD2:2024, based on limb circumference range):

  * Adult Small (19-27 cm) = 165*[8/(2*24)] = 28
  * Adult (25-34 cm) = 165*[9/(2*24)] = 31
  * Adult Large Short (30-40 cm with severely conical arm) = 165*[10/(2*24)] = 35
  * Adult Large (32-43 cm) = 165*[11/(2*24)] = 38
* At least 40% of the subjects within each cuff size shall have a limb circumference that lies within the upper half of the specified range of use of the cuff
* At least 40% of the subjects within each cuff size shall have a limb circumference within the lower half of the specified range of use of the cuff
* At least 10% SBP measurements ≤ 100 mmHg
* At least 10% SBP measurements ≥ 160 mmHg
* At least 10% DBP measurements ≤ 70 mmHg
* At least 10% DBP measurements ≥ 85 mmHg

Exclusion Criteria:

* Emergency surgery
* Surgeries in which both arms are tucked
* Inability to place the Philips AMC appropriately due to subject anatomy or condition
* Known pregnancy or lactating women (self-report)
* Patients treated with an intra-aortic balloon pump
* Aortic and mitral regurgitation (> 2nd degree), if known
* Measurements taken in the lateral position
* Pressure of the arterial line system, when tested at 100 mmHg with the VeriCal device, exceeds the +/- 2 mmHg threshold
* Currently participating in an investigational drug or another device study that clinically interferes with the study endpoints
* Upper arm circumference < 19 cm or > 43 cm
* BMI > 45
* If the average of 3 baseline NIBP lateral difference measurements for SBP is > 15 mmHg or for DBP is > 10 mmHg
* At the PI's discretion, subject does not qualify to participate in the study for any reasons that are not mentioned above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 205 non-cardiac surgical or Intensive Care Unit (ICU) patients being monitored with a radial arterial line will be enrolled over approximately 8 months accrual and follow-up evaluation period.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | Approximately 8 months accrual and follow-up evaluation period.
  The comparison of systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean arterial pressure (MAP) between the Philips AMC and radial arterial line.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University Health System, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
- LMU Klinikum, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No